CLINICAL TRIAL: NCT00349908
Title: A Feasibility Study of the Cordis Neurovascular Self Expanding Stent System in Intracranial Arteries
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Codman & Shurtleff (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CNV:ARG:P-01
Record Dates: First submitted 2006-07-06; First posted 2006-07-10 (Estimated); Results first posted 2013-10-11 (Estimated); Last update posted 2014-06-30 (Estimated); Status verified 2014-05

CONDITIONS: Atherosclerosis; Aneurysm
Keywords: Atherosclerosis,Wide Neck Aneurysm
MeSH Terms: conditions — Atherosclerosis; Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1: Atherosclerosis Arm (Experimental): Implant of Cordis Neurovascular ENTERPRISE Self Expanding Stent System
  Interventions: Device: Cordis Neurovascular ENTERPRISE Self Expanding Stent System
- Group 2: Aneurysm Arm (Active Comparator): Implant of Cordis Neurovascular ENTERPRISE Self Expanding Stent System
  Interventions: Device: Cordis Neurovascular ENTERPRISE Self Expanding Stent System

INTERVENTIONS:
Device: Cordis Neurovascular ENTERPRISE Self Expanding Stent System — Implantation of the device ENTERPRISE used to treat symptomatic stenosis in intracranial arteries.
  Other Names: Other Names:; ENTERPRISE Vascular Reconstruction Device (VRD); ENTERPRISE VRD; ENTERPRISE
  Arms: Group 1: Atherosclerosis Arm
Device: Cordis Neurovascular ENTERPRISE Self Expanding Stent System — Implantation of the device ENTERPRISE to treat wide-necked aneurysms
  Other Names: ENTERPRISE Vascular Reconstruction Device (VRD); ENTERPRISE VRD; ENTERPRISE
  Arms: Group 2: Aneurysm Arm

SUMMARY:
Feasibility study to assess safety of treating patients with self expanding stent in intracranial arteries.

DETAILED DESCRIPTION:
Feasibility study to assess safety of treating patients with self expanding stent in intracranial arteries. Patients will be followed for 6 months with assessments related to technical feasibility and adverse events.

ELIGIBILITY:
Contact site for specific information

Inclusion Criteria:

* Subject meet specific criteria for treatment
* Subject must be willing to return to site for 30 day and 6 month follow up evaluations

Exclusion Criteria:

* Stenting, angioplasty or endarterectomy of an extracranial (carotid or vertebral artery) or intracranial artery within 30 days prior to expected enrollment date
* Previously implanted carotid stent associated with the symptomatic distribution within the past 12 weeks

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-09; Primary Completion 2008-10 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Lylyk, MD, Principal Investigator — ENERI-CLINICA ADVENTISTA BELGRANO
Locations (1):
- Eneri-Clinica Adventista Belgrano, Belgrano, Argentina

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at 1 hospital in Argentina in 2006 and 2007 and treated with Codman Neurovascular Self-Expanding Stent System.
Pre-assignment Details: This is a device study, there was no wash out or run-in phase for transition.
Groups:
- Aneurysm Arm: Intracranial wide-necked aneurysms
- Atherosclerosis Arm: Symptomatic stenosis in intracranial arteries
Period: Overall Study
Arm/Group | Aneurysm Arm | Atherosclerosis Arm
Started | 10 | 10
Completed | 10 | 6 (9 returned for 30 day follow-up, 7 returned for 6 month and 6/7 had 6 month angiogram)
Not Completed | 0 | 4
Not completed — Withdrawal by Subject | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aneurysm Arm | Atherosclerosis Arm | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 9 | 19
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (9.0) | 63.7 (9) | 63.85 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 8 | 8 | 16
Region of Enrollment [Number; unit: participants]
  Argentina | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Technical Feasibility- Successful Stent/Coil Placement (Post Procedure)
Description: Successful placement of the product assessed immediately post procedure
Time Frame: post procedure
Measure: Number; unit: percentage of stable placement
Groups:
- Group 1: Atherosclerosis Arm
- Group 2: Aneurysm Arm
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 10 | 10
percentage of stable placement | 100 (47.3) [0 to 100] | 90 (14.7) [0 to 100]

2. Secondary Outcome: The Secondary Outcome Measure in Group 1, Atherosclerosis and in Group 2, Aneurysm, is the Evaluation of Adverse Events. The Groups Were Analyzed Separately.
Description: An adverse event was defined as any untoward medical occurrence in a subject.
Time Frame: 6 months
Population: Group 1 and Group 2 were analyzed separately. In group 1 Atherosclerosis, 25 unique adverse events were reported in 8 of the 10 eligible subjects. In group 2 aneurysm, 28 unique adverse events were reported in 9 of the 10 eligible subjects.
Measure: Number; unit: Number of adverse events
Groups:
- Group 1: Atherosclerosis
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 10 | 10
Number of adverse events | 25 | 28

3. Primary Outcome: Technical Feasibility- Percent Occlusion (Post Procedure)
Description: Occlusion evaluated immediately post procedure
Time Frame: post procedure
Population: Group 1 - Atherosclerosis Arm not analyzed for occlusion. Occlusion only relevant in Aneurysm treatment.
Measure: Mean (Full Range); unit: percent occlusion
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 0 | 10
percent occlusion |  | 86.8 [0 to 100]

4. Primary Outcome: Technical Feasibility- Percent Occlusion (6 Mo Post Procedure)
Description: 6 Months post
Time Frame: 6 mo
Population: Group 1 - Atherosclerosis Arm not analyzed for occlusion. Occlusion only relevant in Aneurysm treatment.
Measure: Mean (Full Range); unit: percent occlusion
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 0 | 10
percent occlusion |  | 88.8 [0 to 100]

5. Primary Outcome: Technical Feasibility- Successful Stent/Coil Placement (6 Mo Post Procedure)
Description: Successful stent/coil placement assessed at 6 mo post
Time Frame: 6 mo
Measure: Number; unit: Percentage of stable stent/coil placemen
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 10 | 10
Percentage of stable stent/coil placemen | 100 | 100

6. Primary Outcome: Technical Feasibility- Percent Stenosis (6 mo Post Procedure)
Description: Percent Stenosis assessed 6 mo Post Procedure from pre-procedure
Time Frame: 6 mo
Population: Group 2 - Aneurysm Arm not analyzed for stenosis. Stenosis only relevant in Atherosclerosis treatment.
Measure: Mean (Standard Deviation); unit: Percentage change from PreProcedure
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 6 | 0
Percentage change from PreProcedure | -47.3 (21.2) |

7. Primary Outcome: Technical Feasibility- Percent Stenosis (Post Procedure)
Description: Percent Stenosis assessed immediately post procedure from pre procedure
Time Frame: Post Procedure
Population: Group 2 - Aneurysm Arm not analyzed for stenosis. Stenosis only relevant in Atherosclerosis treatment.
Measure: Mean (Standard Deviation); unit: Percentage Change from PreProcedure
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 10 | 0
Percentage Change from PreProcedure | -38.5 (18.3) |

ADVERSE EVENTS:
Time Frame: From the time the informed consent was signed, AEs were assessed after the procedure, at discharge, at thirty days and six months after treatment.
Description: For all enrolled subjects, incidence of AEs assessed immediately following the pre-procedure angiogram through hospital discharge. For subjects with a deployed stent, incidence of AEs assessed immediately following the pre-procedure angiogram through hospital discharge, at thirty days and six months after treatment.
Groups:
- Group 1: Atherosclerosis Arm: This is the events from the Atherosclerosis Arm
- Group 2: Aneurysm Arm: This is the events from the Aneurysm Arm
Arm/Group | Group 1: Atherosclerosis Arm | Group 2: Aneurysm Arm
Serious Adverse Events (participants affected / at risk) | 3/10 | 3/10
Other Adverse Events (participants affected / at risk) | 8/10 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Group 1: Atherosclerosis Arm (N=10) | Group 2: Aneurysm Arm (N=10)
Myocardial Infarction (Cardiac disorders) | 1/1 (1) | 0 (0)
Lung Tumor (Respiratory, thoracic and mediastinal disorders) | 1/1 (1) | 0 (0)
Ischemic Stroke (Nervous system disorders) | 1/1 (1) | 0 (0)
Hip Fracture (Musculoskeletal and connective tissue disorders) | 1/1 (1) | 0 (0)
Stroke/CVA: Ischemic stroke (Nervous system disorders) | 1/1 (1) | 0 (0)
Other: Primitive Left Carotid Ligation (Vascular disorders) | 0 (0) | 1 (1)
Neurological Deficit: left hemianes-thesia and cranial nerve X1 palsy (Vascular disorders) | 0 (0) | 1 (1)
Other: Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Atherosclerosis Arm (N=10) | Group 2: Aneurysm Arm (N=10)
Headache (Nervous system disorders) | 3 (3) | 8 (8)
Hematoma (Nervous system disorders) | 1 (1) | 1 (1)
Hypo-Hypertension (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Ischemia (Nervous system disorders) | 1 (1) | 0 (0)
Myocardial Infarction (Nervous system disorders) | 1 (1) | 0 (0)
Stroke/CVA (Nervous system disorders) | 1 (1) | 0 (0)
Other: Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Other: Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Other: Confusion (Nervous system disorders) | 1 (1) | 1 (1)
Other: Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Other: Elevated Blood Glucose (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Other: Hip Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Other: Insomnia (General disorders) | 1 (1) | 0 (0)
Other: Lung Tumor (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Other: Nausea (General disorders) | 2 (2) | 1 (1)
Other: Postural Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Other: Psychomotor excitation (Nervous system disorders) | 1 (1) | 0 (0)
Other: Tiredness (General disorders) | 1 (1) | 0 (0)
Other: Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1)
Hematoma (Vascular disorders) | 1 (1) | 1 (1)
Hemorrhage (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neurological Deficit (Vascular disorders) | 0 (0) | 2 (2)
Seizures (Vascular disorders) | 0 (0) | 1 (1)
Stent Migration/Embolization (Vascular disorders) | 0 (0) | 1 (1)
Other: Cervical, Dorsal, and/or Lumbar Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Other: Eye Pain Sensation (Eye disorders) | 0 (0) | 1 (1)
Other: Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Other: Photophoby (Eye disorders) | 0 (0) | 1 (1)
Other: Polyuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Other: Primitive Left Carotid Ligation (Vascular disorders) | 0 (0) | 1 (1)
Other: Vomiting (General disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less